CLINICAL TRIAL: NCT07268742
Title: Free Fraction Vitamin D Measurements to Improve Understanding of Steroid Metabolism in Endocrine Disorders
Brief Title: Free Vitamin D and Steroid Metabolism in Endocrine Disorders
Acronym: FREEDOM
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Principal Investigator, Leen Antonio, Prof. Dr., Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S67385
Record Dates: First submitted 2025-11-21; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Vitamin D; Vitamin D and Calcium Homeostasis
Keywords: Vitamin D; Free vitamin D; Free hormone hypothesis
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sampling by venous blood draw;
  * Plasma
  * Serum
  * EDTA-whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Healthy Controls: 1. 264 individuals, consisting of;
     * 132 men
     * 132 women
  2. Intervention - Single venous blood draw
  Interventions: Other: Blood draw for the laboratory assessment
- Obesity: 1. 132 individuals with obesity, subgrouped according to obesity class
     * 33 individuals with overweight, BMI 25.0-29.9 kg/m²
     * 33 individuals in obesity class I BMI 30.0-34.9 kg/m²
     * 33 individuals in obesity class II BMI 35.0-39.9 kg/m²
     * 33 individuals in obesity class III BMI equal to or greater than 40.0 kg/m²
  2. Intervention - Single venous blood draw
  Interventions: Other: Blood draw for the laboratory assessment
- Chronic Kidney Disease: 1. 132 individuals with chronic kidney disease (CKD), subgrouped according to CKD staging;
     * 33 individuals in class 3a, eGFR 45 - 59 mL/min/1.73m²
     * 33 individuals in class 3b, eGFR 30 - 44 mL/min/1.73m²
     * 33 individuals in class 4, eGFR 15 - 29 mL/min/1.73m²
     * 33 individuals in class 5, eGFR <15 mL/min/1.73m²
  2. Intervention - Single venous blood draw
  Interventions: Other: Blood draw for the laboratory assessment
- Pregnancy: 1. 132 pregnant women;
     - recruited during the first trimester of pregnancy
  2. Intervention
     * Venous blood draw
     * At 4 timepoints: trimester 1 (week 1-12) , trimester 2 (week 13-27), trimester 3 (week 28-40) and 4-6 weeks after delivery
  Interventions: Other: Blood draw for the laboratory assessment
- Primary Hyperparathyroidism: 1. 220 individuals with primary hyperparathyroidism
     * New diagnosis or previously untreated by surgery
     * With an indication for surgery (parathyroidectomy, PTX))
  2. Intervention
     * Venous blood draw
     * At 3 timepoints: at diagnosis (pre-PTX), day 1 after PTX and post-PTX (during a standard-of-care follow-up visit)
  Interventions: Other: Blood draw for the laboratory assessment
- Complex calcium/phosphate disorders: 1. Individuals with complex calcium and phosphate homeostasis disorders
  2. Intervention - Single venous blood draw
  Interventions: Other: Blood draw for the laboratory assessment

INTERVENTIONS:
Other: Blood draw for the laboratory assessment — Blood draw for the laboratory assessment

SUMMARY:
This clinical study aims to gain a better understanding of how different forms of vitamin D are processed in the body in healthy individuals, pregnant women, and patients with various hormonal (endocrine) and kidney (renal) disorders. In the long term, this study may provide new insights that could how vitamin D is tested and interpreted in these groups.

Vitamin D has several important roles in the body, such as building strong bones and maintaining calcium balance in the blood. Most vitamin D in the blood circulation is attached/bound to a protein called "vitamin D binding protein" (VDBP), which makes it unavailable for the body to use. A much smaller portion circulates freely in the blood and this is called "free vitamin D". This free form can be directly used by the body.

When your doctor tests your vitamin D levels, this usually refers to total vitamin D (the sum of bound and free vitamin D). However, this total value may not give an accurate indication of your actual vitamin D status, since most of it (the bound part) cannot be used by the body. The purpose of this study is to examine whether "free vitamin D" is a better marker of vitamin D status and if the amount of free vitamin D differs between healthy people, pregnant women, and people with specific endocrine or kidney disorders.

Additionally, this study will look into vitamin D metabolism more detailed, and investigate what different forms of vitamin D exist, how the body processes these, and whether these forms may be related to certain endocrine or kidney conditions.

ELIGIBILITY:
1. General inclusion Criteria:

   - 18 years or above
2. General exclusion Criteria:

   * Below 18 years of age
   * Individuals incapable of providing informed consent
3. Cohort inclusion criteria

   * Obesity: BMI ≥ 25 kg/m2
   * Chronic Kidney Disease: ≥ CKD stage 3a (eGFR < 60 mL/min/1.73m2)
   * Pregnancy: in trimester 1 of pregnancy
   * Primary hyperparathyroidism: diagnosis at UZ Leuven and scheduled for parathyroidectomy at UZ Leuven
   * Complex calcium and phosphate disorders: diagnosis at UZ Leuven
4. Cohort exclusion criteria

   * Healthy controls: BMI below 18 kg/m² or above 25 kg/m², pregnancy, chronic kidney disease (independent of staging), primary hyperparathyroidism and vitamin D and/or calcium supplementation
   * Obesity: chronic kidney disease (independent of staging), pregnancy, primary hyperparathyroidism
   * Chronic Kidney Disease: BMI below 18 kg/m² or above 30 kg/m², pregnancy, primary hyperparathyroidism
   * Pregnancy: BMI below 18 kg/m² or above 30 kg/m², chronic kidney disease (independent of staging), primary hyperparathyroidism
   * Primary hyperparathyroidism: BMI below 18 kg/m² or above 30 kg/m², pregnancy, chronic kidney disease (independent of staging), secondary hyperparathyroidism

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Healthy controls: community sample
  * Other cohorts: recruited from UZ Leuven (Academic medical center/tertiairy care center)
Sampling Method: Non-Probability Sample
Enrollment: 930 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Direct measurement of free 25-hydroxyvitamin D3 levels | - Baseline (all cohorts) - Baseline (trimester 1, week 1-12) , trimester 2 (week 13-27), trimester 3 (week 28-40) and 4-6 weeks after delivery (Pregnancy) - Baseline, perioperative and 4-8 weeks after parathyroidectomy (Primary Hyperparathyroidism)
  1) Direct measurement of free 25-hydroxyvitamin D3, reported as concentration levels per cohort;
  * Reported at baseline
  * Reported as change versus healthy control group (all cohorts vs healthy control)
  * Reported as change within-cohort (Pregnancy and Primary Hyperparathyroidism).

SECONDARY OUTCOMES:
Calculation of free 25-hydroxyvitamin D3 levels | - Baseline (all cohorts) - Baseline (trimester 1, week 1-12) , trimester 2 (week 13-27), trimester 3 (week 28-40) and 4-6 weeks after delivery (Pregnancy) - Baseline, perioperative and 4-8 weeks after parathyroidectomy (Primary Hyperparathyroidism)
  1) Calculation of free 25-hydroxyvitamin D3, reported as concentration levels per cohort;
  * Reported at baseline
  * Reported as change versus healthy control group (all cohorts vs healthy control)
  * Reported as change within-cohort (Pregnancy and Primary Hyperparathyroidism).
Correlation of measured and calculated free 25-hydroxyvitamin D3 levels | - Baseline (all cohorts) - Baseline (trimester 1, week 1-12) , trimester 2 (week 13-27), trimester 3 (week 28-40) and 4-6 weeks after delivery (Pregnancy) - Baseline, perioperative and 4-8 weeks after parathyroidectomy (Primary Hyperparathyroidism)
  Assessment of correlation between measured (Primary Outcome) and calculated (Secondary Outcome 1) free 25-hydroxyvitamin D3 levels
Laboratory assessment of vitamin D metabolite profile | - Baseline (all cohorts) - Baseline (trimester 1, week 1-12) , trimester 2 (week 13-27), trimester 3 (week 28-40) and 4-6 weeks after delivery (Pregnancy) - Baseline, perioperative and 4-8 weeks after parathyroidectomy (Primary Hyperparathyroidism)
  Laboratory assessment of different vitamin D metabolites;
  * 25-hydroxyvitamin D3
  * 3-epi-hydroxyvitamin D3
  * 1(alpha).25-dihydroxyvitamin D3
  * 1(beta).25-dihydroxyvitamin D3
  * 3-epi-1.25-dihydroxyvitamin D3
  * 24.25-dihydroxyvitamin D3
  * 25-hydroxyvitamin D2
  * 1.25-dihydroxyvitamin D2

CONTACTS AND LOCATIONS:
Overall Officials: Leen Antonio, MD, PhD, Principal Investigator — University Hospitals Leuven, Department of Endocrinology
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No